CLINICAL TRIAL: NCT07259252
Title: Influenza Vaccination After Acute Coronary Syndrome
Acronym: InVaACS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tongji Hospital (Other)
Responsible Party: Principal Investigator, Dao Wen Wang, Professor, Tongji Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: InVaACS
Record Dates: First submitted 2025-11-21; First posted 2025-12-02 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Acute Coronary Syndromes (ACS)
MeSH Terms: conditions — Acute Coronary Syndrome | interventions — Influenza Vaccines

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- influenza vaccination (Experimental): patients will receive influenza vaccination
  Interventions: Drug: Influenza vaccine
- placebo (Placebo Comparator): patients will receive placebo (PBS)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Influenza vaccine — Patients receive injection of 0.5ml influenza vaccine
  Arms: influenza vaccination
Drug: Placebo — Patients will receive injection of 0.5ml PBS
  Arms: placebo

SUMMARY:
The goal of this clinical trial is to learn if influenza vaccination can prevent adverse cardiac events in Chinese acute coronary syndrome patients. The main questions it aims to answer are:

* Whether influenza vaccination can decrease events of cardiovascular death, MI, or stroke?
* Whether influenza vaccination can decrease events of all cause death, unplanned revascularization, unplanned hospitalization for heart failure or for arrhythmia, stent thrombosis?

If there is a comparison group: Researchers will compare influenza vaccination and placebo to see if adverse cardiac events decrease.

Participants will receive an influenza vaccination or placebo after enrollment and phone calls for follow-up at 1 month, 3 months, 6 months and 1 year after discharge.

ELIGIBILITY:
Inclusion Criteria:

1. ACS patient aged from 18 to 80 years.
2. Volunteer for the study and written informed consent.

Exclusion Criteria:

1. Participate in any drug clinical trials within 3 months.
2. Patients with life-threatening complications, or the researchers determined that the survival time of patients with no more than 1 years.
3. Serious neurological disease (Alzheimer's disease, Parkinson syndrome, progressive lower limbs or deaf patients).
4. Previous history of cancer or tumor, or pathological examination confirmed precancerous lesions (such as breast ductal carcinoma in situ, or atypical hyperplasia of the cervix).
5. Patients refused to comply with the requirements of this study to complete the research work.
6. Patients Received influenza vaccination within 1 year.
7. Patients with contraindications for influenza vaccination.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6620 (Estimated)
Dates: Start 2025-12-03 (Actual); Primary Completion 2029-03-30 (Estimated); Study Completion 2029-03-30 (Estimated)

PRIMARY OUTCOMES:
Composite endpoint of cardiovascular death, myocardial infarction or stroke | 12 months
  The number of participants with cardiovascular death, myocardial infarction or stroke (first occurring) till 12 months.

SECONDARY OUTCOMES:
all cause death | 12 months
  The number of participants with all cause death till 12 months
cardiovascular death | 12 months
  The number of participants with cardiovascular death till 12 months
stroke | 12 months
  The number of participants with stroke till 12 months
myocardial infarction | 12 months
  The number of participants with myocardial infarction till 12 months
unplanned hospitalization for heart failure or for arrhythmia | 12 months
  The number of participants with unplanned hospitalization for heart failure or for arrhythmia till 12 months
unplanned revascularization | 12 months
  The number of participants with unplanned revascularization till 12 months
stent thrombosis | 12 months
  The number of participants with stent thrombosis till 12 months

OTHER OUTCOMES:
influenza like illness | 12 months
  The number of participants with fever (body temperature ≥38℃) accompanied by cough or sore throat till 12 months
hospitalization for influenza | 12 months
  The number of participants with hospitalization for influenza till 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Dao Wen Wang, Principal Investigator — Tongji Hospital
Locations (1):
- Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No